CLINICAL TRIAL: NCT06113250
Title: Effect of Shortwave Diathermy Versus Ultrasound Waves on Increasing Rom and Decreasing Pain After Extensor Tendon Reconstruction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ibrahim Yousef Zidane, Lecturer of physical therapy for integumentary disorders, faculty of physical therapy, kafrelsheikh university, Kafrelsheikh University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-29
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Extensor Tendon Reconstruction
Keywords: shortwave diathermy, ultrasound waves, extensor tendon reconstruction, pain, ROM, visual analque scale, goniometer
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: 60 male and female patients will participate in the study are divided into 3 groups (20 in each group). They will be randomly assigned to three equal groups: Group (A): twenty patients will receive shortwave diathermy and traditional physical therapy program (splinting, stretching exercises, strengthening exercises and range of motion (ROM) exercises).
  Group (B): twenty patients will receive ultrasound waves and traditional physical therapy program (splinting, stretching exercises, strengthening exercises and range of motion (ROM) exercises).
  Group (C): twenty patients will receive only traditional physical therapy program (splinting, stretching exercises, strengthening exercises and range of motion (ROM) exercises)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- shortwave diathermy (Active Comparator)
  Interventions: Device: shortwave diathermy
- ultrasound waves (Active Comparator)
  Interventions: Device: ultrasound waves
- therapeutic exercises (Sham Comparator)
  Interventions: Device: shortwave diathermy; Device: ultrasound waves; Other: traditional physical therapy program

INTERVENTIONS:
Device: shortwave diathermy — Shortwave diathermy (SWD) is a modality that produces heat by converting electromagnetic energy into thermal energy. pulsed shortwave diathermy (PSWD), uses high-frequency electromagnetic waves to heat tissues up to 5 cm deep. Heat is produced by the resistance of tissue to the passage of energy. Although it heats to the same depth as 1-MHz ultrasound, PSWD heats a much larger area than ultrasound does, making it ideal to heat larger joints, such as the elbow, shoulder, hip, knee, and ankle
  Arms: shortwave diathermy; therapeutic exercises
Device: ultrasound waves — Ultrasound is sound with a frequency above 20,000 Hertz (Hz) and is undetectable by the human ear. However, clinical ultrasound uses much high frequencies of between 1 and 20 megahertz (MHz) and sometimes up to 75 MHz in specialized areas such as dermatology and ophthalmology. Clinically, ultrasound is used for a number of applications ranging from visualizing structures to allow safe insertion of lines and catheters to diagnostic imaging including the assessment of the movement of cardiac Production of ultrasound waves is the first part of the clinical ultrasound process. Ultrasound is generated by piezoelectric crystals. These crystalline materials contain randomly oriented electric dipoles, and when a force is applied that deforms the crystal, the dipoles are rearranged and a net charge induced across the crystal
  Arms: therapeutic exercises; ultrasound waves
Other: traditional physical therapy program — splinting, stretching exercises, strengthening exercises and range of motion (ROM) exercises
  Arms: therapeutic exercises

SUMMARY:
tendon injuries can result in long-term sequelae, including chronic pain and mobility restrictions, and may warrant surgery. Ultrasound is sound with a frequency above 20,000 Hertz (Hz) and is undetectable by the human ear. Ultrasound waves are generated by a piezoelectric effect caused by vibration of crystals within the head of the wand/probe. The sound waves that pass through the skin cause vibration of the local tissue. This can cause a deep heating locally. ultrasound can provide several benefits for treating strains, sprains, tissue healing andpain.n Shortwave diathermy is a high frequency current that is obtained by a discharging condenser through inductance of low ohmic resistance. When this high frequency current passes into the tissues, it produces heat into the tissues. PSWD heats a much larger area than ultrasound does, making it ideal to heat larger joints, such as the elbow, shoulder, hip, knee, and ankle. This work aims to compare between the effect of shortwave diathermy versus ultrasound waves on increasing ROM and decreasing pain after extensor tendon reconstruction. Sixty adults patients of both sex, aged from 20 to 30 years, with extensor tendon injuries participated in this study after reconstruction surgeries. They were randomly categorized into three groups of equal numbers. Group A received Pulsed shortwave diathermy and traditional physical therapy program (splinting, stretching exercises, strengthening exercises and range of motion (ROM) exercises), group B received ultrasound waves and traditional physical therapy program (splinting, stretching exercises, strengthening exercises and range of motion (ROM) exercises, while group C received only traditional physical therapy program (splinting, stretching exercises, strengthening exercises and range of motion (ROM) exercises). Pain and finger flexion range of motion will be measured before and after two months of intervention. Data and results will be statistically analyzed to give conclusions

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 20 to 30 years
2. After extensor tendon reconstruction surgeries
3. Gender: both male and female

Exclusion Criteria:

1. Photosensitivity
2. Sensory impairements
3. Intellectual disorders
4. Pregnant women

Ages: 22 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-07 (Estimated)

PRIMARY OUTCOMES:
pain at extensor tendons | pain is measured before starting study and after 2 months of intervention
  visual analque scale is a 10 point line is used to quantify amount of pain at extensor tendon of hand
finger flexion ROM | flexion range of finger is measured before starting study and after 2 months
  goniometer is digital tool is used to measure range of finger flexion of hand

CONTACTS AND LOCATIONS:
Overall Officials: Abdelaziz A sherif, Principal Investigator — Vice Dean for graduate studies and research
Locations (1):
- Faculty of Physical Therapy, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt